CLINICAL TRIAL: NCT03010904
Title: The Effect of Pasteurized; Pasteurized and Homogenized and UHT -Treated Homogenized Cow's Milk on Gastrointestinal Symptoms in Sensitive Adults
Brief Title: The Effect of Pasteurized; Pasteurized and Homogenized and UHT Treated Homogenized Cow's Milk on Gastrointestinal Symptoms in Sensitive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Principal investigator, University of Turku
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MILK2
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Unidentified Gastrointestinal Discomfort Following Dairy Consumption
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- pasteurized milk (Experimental): milk that has undergone pasteurization treatment
  Interventions: Other: Dietary intervention
- homogenized pasteurized milk (Experimental): Milk that has undergone homogenization and pasteurization treatment
  Interventions: Other: Dietary intervention
- UHT milk (Experimental): Milk that has undergone homogenization and ultra high temperature treatment
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention

SUMMARY:
This study aims to investigate differences in digestion rates and gastrointestinal problems caused by pasteurized; pasturized and homogenized as well as UHT-treated homogenized cow's milks in healthy adults by diary of symptoms, blood glucose and triacylglycerol levels and plasma cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Homogenized and pasteurized milk causes gastrointestinal problems (self-reported) unhomogenized and unpasteurized milk does not cause gastrointestinal problems (self-reported)
* age 18-65
* BMI 18,5 - 30
* hemoglobin under normal range
* fasting plasma alanine aminotransferase ALAT < 60 U/l (normal liver function)
* fasting plasma thyroid-stimulating hormone (TSH) 0.4 - 4.5 mU/l (normal thyroid function)
* fasting plasma creatinine < 118 umol/l (normal kidney function)

Exclusion Criteria:

* pace maker
* Crohn's disease or other disease of the intestinal tract
* intestinal operation within the last 3 months
* difficult dysphagia
* smoking
* constipation
* lactose intolerance
* coeliac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms (self reported) | day 0 - day 5
  Gastrointestinal symptoms (self-reported) as measured by a questionnaire. The questionnaire is devided into seven types of gastrointestinal discomfort, and also includes a possibility to describe a gastrointestinal discomfort outside these seven given alternatives. The severity of the symptoms is self-reported on a three-step scale.

SECONDARY OUTCOMES:
Plasma triacylglycerols | 20 min, 40 min, 60 min, 120 min, 180 min, 240 min, 300 min
Plasma glucose | 20 min, 40 min, 60 min, 120 min, 180 min, 240 min, 300 min
Plasma insulin | 20 min, 40 min, 60 min, 120 min, 180 min, 240 min, 300 min

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa M Linderborg, PhD, Principal Investigator — Department of Biochemistry, University of Turku
Locations (2):
- Finland (2):
  - Department of Biochemistry, University of Turku, Turku
  - Food Chemistry, Department of Biochemistry, University of Turku, Turku